CLINICAL TRIAL: NCT01321385
Title: Validation of a Classifier for Induction Response Prediction Using Single Cell Network Profiling (SCNP) Assays for Childhood AML
Brief Title: Biomarkers in Predicting Response to Treatment in Bone Marrow Samples From Young Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML11B8; COG-AAML11B8 (Other: Children's Oncology Group); NCI-2011-02851 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AAML11B8 (Other: Children's Oncology Group)
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; childhood acute erythroleukemia (M6); childhood acute megakaryocytic leukemia (M7); childhood acute monoblastic leukemia (M5a); childhood acute monocytic leukemia (M5b); childhood acute myeloblastic leukemia with maturation (M2); childhood acute myeloblastic leukemia without maturation (M1); childhood acute myelomonocytic leukemia (M4); childhood acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — bone marrow
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: laboratory biomarker analysis
Other: study of socioeconomic and demographic variables

SUMMARY:
RATIONALE: Studying samples of bone marrow from patients with cancer in the laboratory may help doctors predict how well patients will respond to treatment.

PURPOSE: This research trial is studying biomarkers in predicting response to treatment in bone marrow samples from young patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To validate the accuracy of a pre-specified acute myeloid leukemia (AML) induction response classifier or the My Profile™ AML Induction Therapy Assay (run in a Good Laboratory Practice [GLP] laboratory using Good Manufacturing Practice [GMP] reagents) in predicting response to cytarabine-based induction chemotherapy in pediatric patients with non-M3 AML.

Secondary

* To validate the continuous score from the pre-specified induction response classifier as a predictor of response to induction chemotherapy, after controlling for the simultaneous effects of clinical variables at base-line and/or pre-induction therapy (e.g., age, WBC, and percentage [%] of blasts), and tests commonly available after the start of induction therapy (e.g., cytogenetics and molecular markers).
* To validate the accuracy of the pre-specified induction response classifier as a binary predictor of induction response using a pre-specified cutpoint to assign patients to no response (NR) or complete response (CR) groups.
* To validate the accuracy of the pre-specified induction response classifier as a binary predictor of induction response using a pre-specified cutpoint to assign patients to NR or CR groups, after controlling for the simultaneous effects of clinical variables at base-line (pre-induction therapy) (e.g., age, WBC, % blasts) and clinical variables, including tests commonly available after start of induction therapy (e.g., age, WBC, cytogenetics).

OUTLINE: Cryopreserved bone marrow mononuclear cell specimens are analyzed by cell networking profiling assays. Results are then compared with patient outcomes and demographics from COG-AAML03P1 and COG-AAML0531 studies.

Molecular markers analyzed include Flt3ITD, NPM1, CEBPA, and MRA.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML)

  * Non-M3 AML
* Cryopreserved bone marrow mononuclear cell specimens from patients enrolled on COG-AAML03P1 and COG-AAML0531 collected prior to cytarabine-based induction therapy

  * Patient samples from COG-AAML0531 must come from the control arm (i.e., no gemtuzumab ozogamicin induction therapy)

PATIENT CHARACTERISTICS:

* No Down syndrome

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosis of acute myeloid leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2011-03; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Accuracy of induction response prediction

SECONDARY OUTCOMES:
Duration of complete response
Event-free survival and overall survival
Status (dead vs living)
Date of last follow up

CONTACTS AND LOCATIONS:
Overall Officials: Norman J. Lacayo, MD, Principal Investigator — Stanford University